CLINICAL TRIAL: NCT06888856
Title: Observational Study on Genomic and Proteomic Mechanisms in Multiple Myeloma Patients Treated With Bispecific Antibodies and CAR-T Therapies
Brief Title: Multiple Myeloma is a Hematologic Malignancy Characterized by the Accumulation of Malignant Plasma Cells in the Bone Marrow. Despite Advances in Treatment, Many Patients Experience Disease Relapse. Bispecific Antibodies Offer an Innovative Therapeutic Approach, But Approximately 30%-40% of Patients
Acronym: MMOMICS
Status: Not yet recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0523-24 TLV; 0523-24 TLV (Registry Identifier: MMOMICS)
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Bone Marrow, Serum, Peripheral Blood Mononuclear Cells (PBMCs), Plasma Cells (CD138+) These samples will be used for various analyses including flow cytometry, ELISA (for soluble BCMA), single-cell RNA sequencing, and genomic DNA sequencing of specific regions from myeloma cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, non-interventional study aims to characterize the molecular and cellular mechanisms underlying the response and resistance of multiple myeloma (MM) patients to bispecific antibodies (BisAb) and CAR-T therapies. Conducted at the Tel Aviv Sourasky Medical Center, the study will enroll up to 200 MM patients aged 18 and older, who are candidates for BisAb, CAR-T, or other MM treatments. Bone marrow (4-6 mL) and peripheral blood (15-20 mL) samples will be collected before treatment and at predefined intervals post-treatment, including at disease relapse/progression. The study will analyze plasma cells and the tumor microenvironment (TME) using techniques such as flow cytometry (FACS), single-cell RNA sequencing, genomic DNA sequencing, and ELISA to assess soluble BCMA levels. Key objectives include identifying genetic and protein signatures predictive of treatment response, evaluating specific drug binding, and analyzing interactions between plasma cells and immune cells (e.g., T cells). Samples will be processed and stored at the study site, with data coded to ensure patient confidentiality. Results will inform personalized treatment strategies for MM patients. The study duration includes 5 years for sample collection, 1 year for data analysis, and up to 20 years for sample storage.

DETAILED DESCRIPTION:
The study protocol outlines a prospective, non-interventional research initiative at Tel Aviv Sourasky Medical Center to investigate molecular mechanisms of response and resistance to bispecific antibodies (BisAb) and CAR-T therapies in multiple myeloma (MM) patients. Led by Prof. Yael Cohen, the study aims to personalize treatment by analyzing bone marrow (4-6 mL) and peripheral blood (15-20 mL) samples from up to 200 MM patients aged 18+, collected pre-treatment and at specific post-treatment intervals (e.g., relapse). Key methods include flow cytometry (FACS) for drug binding and cell interactions, single-cell RNA sequencing and genomic DNA sequencing for genetic profiling, and ELISA for soluble BCMA levels. Plasma cells and the tumor microenvironment (TME) will be characterized to identify predictive biomarkers, focusing on genes like BCMA, GPRC5D, and FcRL5. Samples will be processed and stored at the study site for up to 20 years, with strict confidentiality ensured through coding. The study spans 5 years for sample collection, 1 year for analysis, and aims to improve MM treatment outcomes through tailored therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with multiple myeloma Candidate for BisAb, CAR-T, or other myeloma therapy Mentally competent and able to sign informed consent

Exclusion Criteria:

Unable to undergo bone marrow sampling Pregnant women Minors (<18), incapacitated, or legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of up to 200 adults diagnosed with Multiple Myeloma who are receiving or have received bispecific antibodies or CAR-T therapies. Participants will provide bone marrow and blood samples to study treatment response and resistance mechanisms. Participants must consent to data collection regarding their disease and treatment history.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-19 (Estimated); Primary Completion 2030-03-03 (Estimated); Study Completion 2031-03-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between molecular/cellular characteristics and treatment response | Up to 5 years (duration of sample collection) plus 1 year for analysis
  Assessment of correlation between pre-treatment molecular and cellular characteristics (including specific drug binding, plasma cell-T cell interactions, gene expression profiles, genomic mutations in therapeutic targets, and soluble BCMA levels) and clinical response to bispecific antibody and CAR-T cell therapies in multiple myeloma patients. Samples will be collected before treatment initiation and at fixed timepoints after treatment begins, with response evaluated according to standard multiple myeloma response criteria

IPD SHARING:
Plan to Share IPD: No
No individual patient data (IPD) will be shared outside the hospital. All data will be securely coded and stored within the hospital's internal systems with limited access, ensuring the confidentiality and privacy of participants.